CLINICAL TRIAL: NCT06846437
Title: A Randomized, Controlled, Open-Label, Multicenter, Phase 3 Study to Compare the Efficacy and Safety of JSKN003 Versus Trastuzumab Emtansine (T-DM1) for HER2-Positive, Advanced Breast Cancer Subjects
Brief Title: JSKN003 Versus Trastuzumab Emtansine (T-DM1) for HER2-Positive, Advanced Breast Cancer
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Shanghai JMT-Bio Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: JSKN003-301
Record Dates: First submitted 2025-01-06; First posted 2025-02-26 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2025-02

CONDITIONS: Unrespectable Locally Advanced and or Metastatic HER2 Positive Breast Cancer Participants
MeSH Terms: interventions — Ado-Trastuzumab Emtansine

STUDY DESIGN:
Intervention Model Description: This is a randomized, controlled, open-label, multicenter, phase 3 clinical study. The primary endpoint of this study is PFS as assessed by BIRC. Participants with unrespectable locally advanced and/or metastatic HER2-positive breast cancer previously treated with trastuzumab and taxane are randomly assigned 1:1 stratified by hormone receptor status (positive or negative) and previous treatment lines (1L or ≥2L) to receive JSKN003 (experimental) or T-DM1 (active comparator).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- JSKN003 (Experimental): Received JSKN003 as a sterile intravenous (IV) solution at a dose of 6.3 mg/kg every 3 weeks (Q3W).
  Interventions: Drug: JSKN003
- T-DM1 (Active Comparator): Received T-DM1 in accordance with the approved label.
  Interventions: Drug: Trastuzumab emtansine (T-DM1)

INTERVENTIONS:
Drug: JSKN003 — Administered intravenously according to protocol.
  Arms: JSKN003
Drug: Trastuzumab emtansine (T-DM1) — Administered intravenously according to the approved label.
  Arms: T-DM1

SUMMARY:
This study is designed to compare the safety and efficacy of JSKN003 versus T-DM1 in unrespectable locally advanced and/or metastatic HER2-positive breast cancer participants previously treated with trastuzumab and taxane.

DETAILED DESCRIPTION:
This is a randomized, controlled, open-label, multicenter, phase 3 clinical study to compare the efficacy and safety of JSKN003 versus T-DM1 in unresectable locally advanced and/or metastatic HER2-positive breast cancer participants previously treated with trastuzumab and taxane. Participants will be treated with JSKN003 at 6.3 mg/kg or trastuzumab emtansine at 3.6 mg/kg every 3 weeks (Q3W). Participants will continue to receive treatment until disease progression, intolerable toxicity, withdrawal of informed consent, death, or any other reasons for treatment discontinuation, whichever occurs first.

ELIGIBILITY:
Inclusion Criteria:

* 1. Voluntarily agree to participate in the study and sign the informed consent.
* 2.Age≥18 years old.
* 3.Patients with unresectable locally advanced or metastatic breast cancer confirmed by histology or cytology.
* 4.Confirmed to be HER2 positive (HER2-positive is defined as IHC 3+ or IHC 2+ with ISH positive) by the pathology department of participating study center.
* 5.Have received treatment regimen including trastuzumab (allowed marketed trastuzumab biosimilars) or inetetamab with radiologic or pathologic progression/ relapse during the advanced stage, during neoadjuvant or adjuvant therapy, or within 12 months after treatment.
* 6.Previously treated with taxanes.
* 7.Had radiologic and/or pathologic progression or intolerance of the latest systemic anti-tumor therapy.
* 8.At least one extracranial measurable lesion at baseline according to RECIST 1.1 criteria.
* 9.ECOG PS of 0 - 1.
* 10.Patients with adequate organ and bone marrow functions.
* 11.Expected survival ≥ 3 months.
* 12.Female and male patients of childbearing age agree to take adequate contraceptive measures during and upon completion of the study for 7 months after the last dose of JSKN003 or T-DM1.

Exclusion Criteria:

* 1. Have previously been treated with an anti-HER2 ADC loaded with topoisomerase I inhibitors or medenosin derivative 1 (DM1) or have relapsed after receiving such therapy during or within 12 months after the adjuvant/neo-adjuvant setting or in the advanced stage.
* 2.History of any other malignant tumors within three years before randomization.
* 3.With uncontrollable serous effusion within 14 days before randomization, which requires frequent drainage or medical intervention.
* 4.Known contraindication to T-DM1or not suitable to receive JSKN003 or T-DM1 by investigator.
* 5.Has not recovered from adverse reactions caused by previous anti-tumor treatments to ≤ Grade 1 (refer to NCI CTCAE 5.0) or baseline (excluding grade 2 alopecia, hyperpigmentation, simple laboratory test abnormalities, and other toxicity for a non-safety risk by investigators).
* 6.Received immunotherapy, macromolecular targeted therapy or other anti-tumor biological therapy within 4 weeks before randomization, or received palliative radiotherapy, endocrine therapy, cytotoxic drug chemotherapy and small molecular targeted drug therapy within 2 weeks before randomization, or received traditional Chinese medicine preparations with anti-tumor indications within 2 weeks before randomization.
* 7.Major organ surgery within 28 days before randomization.
* 8.Untreated (including baseline findings) or unstable cerebral parenchymal metastasis, spinal cord metastasis or compression, and cancerous meningitis.
* 9.The cumulative amount of previous exposure to anthracyclines has reached the pre-specified dosage.
* 10.History of LVEF < 40% during prior anti-HER2 drug therapy or symptomatic congestive heart failure (CHF).
* 11.Serious or uncontrolled cardiovascular disease.
* 12.History of (non-infectious) interstitial lung disease/pneumonitis requiring therapy or grade ≥3 interstitial lung disease/ pneumonitis during previous anti-tumor treatments.
* 13.Active infections requiring intravenous antibiotics, antivirals, or antifungals within 14 days before randomization.
* 14. Active hepatitis B or hepatitis C.
* 15.History of immunodeficiency or HIV antibody test positive at screening.
* 16.Received a potent inhibitor of CYP3A4 within 14 days prior to randomization or during study treatment.
* 17.Pregnant or nursing females;
* 18.Other reasons enrolled in this clinical trial as considered unsuitable by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 228 (Estimated)
Dates: Start 2025-02-18 (Actual); Primary Completion 2026-10-13 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival (PFS) by BIRC | Up to approximately 4 years

SECONDARY OUTCOMES:
Progression-free survival (PFS) by investigator | Up to approximately 4 years
Overall Survival (OS) | Up to approximately 4 years
Objective Response Rate (ORR) | Up to approximately 4 years
Disease Control Rate (DCR) | Up to approximately 4 years
Duration of Response (DoR) | Up to approximately 4 years
Incidence and severity of TEAE and SAE | From the signing of informed consent to the safety follow-up period or before starting a new anti-tumor therapy, whichever occurs first, assessed up to approximately 4 years.
Cmax of JSKN003 | Cycles 1, 2, 3, 4 (each cycle is 3 weeks), and every 4 cycles starting from Cycle 4; End of treatment and safety follow-up visit, for approximately 4 years
AUC of JSKN003 | Cycles 1, 2, 3, 4 (each cycle is 3 weeks), and every 4 cycles starting from Cycle 4; End of treatment and safety follow-up visit, for approximately 4 years
Incidence of anti-drug antibodies (ADA) to JSKN003 | Pre-dose for Cycles 1, 2, 3, 4 (each cycle is 3 weeks), and every 4 cycles starting from Cycle 4; End of treatment and safety follow-up visit, for approximately 4 years.

CONTACTS AND LOCATIONS:
Overall Officials: Zhimin Shao, M.D. Organizational Affiliatio, Principal Investigator — Fudan University
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, China